CLINICAL TRIAL: NCT00976300
Title: Cyclosporine A or Intravenous Cyclophosphamide for Lupus Nephritis: The Cyclofa-Lune Study
Acronym: CYCLOFA-LUNE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Rheumatology, Prague (Other)
Collaborators: Ministry of Health, Czech Republic (Other Government); Charles University, Czech Republic (Other); Palacky University (Other); Department of Rheumatology, Hospital, Ceske Budejovice, Czech Republic (Unknown); National Institute of Rheumatology, Piestany, Slovakia (Unknown); St. Anna Hospital, Brno, Czech (Other)
Responsible Party: Institute of Rheumatology, Prague
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RU 8444-3; IGA MZ CR 8444-3; MZO 00023728
Record Dates: First submitted 2009-09-11; First posted 2009-09-14 (Estimated); Last update posted 2010-06-23 (Estimated); Status verified 2009-09

CONDITIONS: Systemic Lupus Erythematosus; Lupus Nephritis
Keywords: SLE; lupus nephritis; cyclosporine A; cyclophosphamide; active proliferative lupus nephritis (class III or IV according to WHO)
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Lupus Nephritis | interventions — Cyclosporine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cyclosporine A (Experimental): Cyclosporine arm (CyA group) consisted of oral cyclosporine A (CyA) 4-5mg/kg/day (given in two divided doses) for 9 months followed by gradually decreasing dose of cyclosporine (3.75-1.25 mg/kg/day) within the next 9 months.
  Interventions: Drug: Cyclosporine A
- Cyclophosphamide (Active Comparator): Cyclophosphamide (CPH) therapeutic arm (CPH group) consisted of 8 boluses of intravenous cyclophosphamide (10mg/kg) given within 9 months in subsequently prolonged intervals (2x3weeks, 4x4 weeks, 2x6 weeks) followed by 4-5 oral cyclophosphamide boluses (10mg/d in 6-8 week intervals).
  Interventions: Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Cyclosporine A — Cyclosporine arm (CyA group) consisted of oral cyclosporine A (CyA) 4-5mg/kg/day (given in two divided doses) for 9 months followed by gradually decreasing dose of cyclosporine (3.75-1.25 mg/kg/day) within the next 9 months. The dosage of concomitant glucocorticoids was driven and tapered according to a single treatment protocol.
  Arms: Cyclosporine A
Drug: Cyclophosphamide — Cyclophosphamide (CPH) therapeutic arm (CPH group) consisted of 8 boluses of intravenous cyclophosphamide (10mg/kg) given within 9 months in subsequently prolonged intervals (2x3weeks, 4x4 weeks, 2x6 weeks) followed by 4-5 oral cyclophosphamide boluses (10mg/d in 6-8 week intervals). The dosage of concomitant glucocorticoids was driven and tapered according to a single treatment protocol.
  Arms: Cyclophosphamide

SUMMARY:
Intravenous cyclophosphamide is considered to be the standard of care for treatment of proliferative lupus nephritis. However, its use is limited by potentially severe toxic effects. Cyclosporine A has been suggested to be an efficient and safe treatment alternative to cyclophosphamide. In a randomized, multicenter, open-label, controlled trial the investigators sought to compare the efficacy of oral cyclosporine A with intravenous pulse cyclophosphamide to induce durable remission in patients with lupus nephritis III-IV.

DETAILED DESCRIPTION:
Lupus nephritis occurs in 30-40% of adults with systemic lupus erythematosus and is associated with increased morbidity and mortality. Focal and diffuse proliferative forms of lupus nephritis are known to progress to chronic renal failure unless treated by immunosuppressive drugs. Cyclophosphamide and glucocorticoids are considered to be the standard of care for patients with proliferative lupus nephritis. However, cyclophosphamide may cause a number of toxic effects, such as bone marrow suppression, premature gonadal failure, hemorrhagic cystitis, opportunistic infections, and malignant disease. Hence, efforts are being made to find alternative therapeutic approaches. Cyclosporine is a potent immunosuppressive agent with a more selective mode of action through its unique effect on T cell mediated responses, and is widely used to treat a spectrum of autoimmune and glomerular diseases. Several retrospective series and one randomized trial provided evidence that Cyclosporine A could represent an efficient and safe therapy for proliferative lupus nephritis. In a randomized, multicenter, open-label, controlled trial we compared the efficacy of oral cyclosporine A with intravenous pulse cyclophosphamide to induce durable remission in patients with proliferative lupus nephritis.

ELIGIBILITY:
Inclusion Criteria:

* the diagnosis of systemic lupus erythematosus (by meeting 4 criteria of the American College of Rheumatology)
* renal biopsy documenting lupus nephritis according to the classification of the World Health Organization (WHO) or the updated International Society of Nephrology/Renal Pathology Society (ISN/RPS) as proliferative glomerulonephritis class III (focal) or IV (diffuse)
* clinical activity as defined by presence of at least two of the following:

  * abnormal proteinuria (more than 500mg of protein in in a 24-hour urine specimen)
  * abnormal microscopic hematuria, or
  * C3 hypocomplementemia (the latter two were defined according to the norms in the laboratories of the participating centers)

Exclusion Criteria:

* treatment with cyclophosphamide or cyclosporine A ever before
* treatment with other immunosuppressive drugs (such as azathioprine or mycophenolate mofetil) or high dose glucocorticoids (≥ 80mg of prednisone or methylprednisolone) within the last 3 months
* persistent elevation of serum creatinine (≥140 μmol/l)
* pregnancy or lactation
* bone marrow insufficiency with cytopenias not attributable to SLE, and 8severe coexisting conditions, such as infection, liver disease, active peptic ulcer etc.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2002-01; Primary Completion 2008-05 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
renal remission and renal response | at the end of induction (month 9) and maintenance (month 18) phase

SECONDARY OUTCOMES:
incidence of adverse events and relapse free period | 18 months

CONTACTS AND LOCATIONS:
Locations (4):
- Czechia (4):
  - Department of Rheumatology, Faculty of Medicine, Charles University in Prague, Hradec Králové
  - Department of Rheumatology, Faculty of Medicine, Palacky University, Olomouc
  - Department of Nephrology, General Teaching Hospital and First faculty of Medicine, Charles University in Prague, Prague
  - Institute of Rheumatology, Prague

REFERENCES:
- [Background] Rihova Z, Vankova Z, Maixnerova D, Dostal C, Jancova E, Honsova E, Merta M, Rysava R, Tesar V. Treatment of lupus nephritis with cyclosporine - an outcome analysis. Kidney Blood Press Res. 2007;30(2):124-8. doi: 10.1159/000101448. Epub 2007 Mar 30. PMID 17396037
- [Background] Dostal C, Tesar V, Rychlik I, Zabka J, Vencovsky J, Bartunkova J, Stejskalova A, Tegzova D. Effect of 1 year cyclosporine A treatment on the activity and renal involvement of systemic lupus erythematosus: a pilot study. Lupus. 1998;7(1):29-36. doi: 10.1191/096120398678919714. PMID 9493146
- [Background] Yee CS, Gordon C, Dostal C, Petera P, Dadoniene J, Griffiths B, Rozman B, Isenberg DA, Sturfelt G, Nived O, Turney JH, Venalis A, Adu D, Smolen JS, Emery P. EULAR randomised controlled trial of pulse cyclophosphamide and methylprednisolone versus continuous cyclophosphamide and prednisolone followed by azathioprine and prednisolone in lupus nephritis. Ann Rheum Dis. 2004 May;63(5):525-9. doi: 10.1136/ard.2002.003574. PMID 15082482
- [Derived] Zavada J, Pesickova S, Rysava R, Olejarova M, Horak P, Hrncir Z, Rychlik I, Havrda M, Vitova J, Lukac J, Rovensky J, Tegzova D, Bohmova J, Zadrazil J, Hana J, Dostal C, Tesar V. Cyclosporine A or intravenous cyclophosphamide for lupus nephritis: the Cyclofa-Lune study. Lupus. 2010 Oct;19(11):1281-9. doi: 10.1177/0961203310371155. Epub 2010 Jul 6. PMID 20605876